CLINICAL TRIAL: NCT06730308
Title: A Prospective, Single-arm Phase II Study of Glucocorticoids Combined With Concurrent Chemoradiotherapy for Unresectable Thymoma
Brief Title: Glucocorticoids Combined With Concurrent Chemoradiotherapy for Unresectable Thymoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GASTO10106
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Thymoma
Keywords: Thymoma; Concurrent chemoradiotherapy; Methylprednisolone
MeSH Terms: conditions — Thymoma | interventions — Radiotherapy; Methylprednisolone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study arm (Experimental): Methylprednisolone combined with concurrent chemoradiotherapy
  Interventions: Radiation: Radiotherapy; Drug: Concurrent chemotherapy; Drug: Methylprednisolone

INTERVENTIONS:
Radiation: Radiotherapy — Hypofractionated radiotherapy
Drug: Concurrent chemotherapy — weekly albumin-bound paclitaxel (50 mg/m²) and cisplatin (25 mg/m²)
Drug: Methylprednisolone — Methylprednisolone 2mg/kg, qd, concurrent with radiotherapy

SUMMARY:
This study aims to assess the efficacy of methylprednisolone combined with concurrent chemoradiotherapy in treating unresectable or recurrent thymoma.

DETAILED DESCRIPTION:
This study aims to assess the efficacy of methylprednisolone combined with concurrent chemoradiotherapy in treating unresectable or recurrent thymoma. Patients will receive hypofractionated radiotherapy with concurrent chemotherapy.

Methylprednisolone will be administered daily during radiotherapy at a dose of 2 mg/kg.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed type AB or B1-3 thymoma.
* Measurable Disease: Patients must have measurable disease as defined by RECIST (Response Evaluation Criteria in Solid Tumors).
* Unresectable or recurrent thymoma, with the tumor confined to the chest and neck area.
* Between the ages of 18 and 70 years, regardless of sex.
* Eastern Cooperative Oncology Group performance status of 0 or 1.
* No prior chest radiation.
* Adequate organ Functions.
* Written informed consent obtained.

Exclusion Criteria:

* Contraindications to Methylprednisolone.
* History of or Concurrent Malignancy.
* Active infection, myocardial infarction within the last 6 months or symptomatic heart disease.
* Pregnant or Lactating Women.
* Bleeding Disorders.
* Recent Participation in Other Clinical Trials.
* Drug Abuse or Severe Alcoholism.
* Uncontrolled Seizures or Mental Disorders.
* Severe Allergies or Specific Sensitivities.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2028-11-19 (Estimated); Study Completion 2028-11-19 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 1-2 months after chemoradiotherapy
  The percentage of patients who achieve complete remission or partial remission after chemoradiotherapy

SECONDARY OUTCOMES:
Progression-free survival | 2-year
  From the start date of initial treatment to progression, death or last follow-up
Overall survival | 2-year
  From the start date of initial treatment to death or to last follow-up.
Toxicities using the CTCAE 5.0 | 1 year after treatment
  Toxicities were evaluated using the CTCAE 5.0
Quality of life scores | 1 year after treatment
  Quality of life assessed by QLQ-C30

CONTACTS AND LOCATIONS:
Locations (1):
- Sun yat-sen University Cancer Center, Guanzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided